CLINICAL TRIAL: NCT01906125
Title: A Phase 1, Open-Label 3 Sequence 3 Period Crossover Study Of Palbociclib (PD-0332991) In Healthy Volunteers To Establish The Bioequivalence Of The Phase 1/2 And Phase 3 Formulation To Palbociclib ICH Formulation Under Fasted Conditions
Brief Title: A Study To Establish The Equivalence Of 2 Palbociclib (PD-0332991) Formulations To The Intended Final Market Product
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A5481020
Record Dates: First submitted 2013-07-16; First posted 2013-07-23 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: Bioequivalence; Cmax; AUC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palbociclib given to Healthy Volunteers (Experimental)
  Interventions: Drug: palbociclib capsule: phase 1 and 2 studies; Drug: Palbociclib capsule: phase 3 studies; Drug: Palbociclib capsule: ICH

INTERVENTIONS:
Drug: palbociclib capsule: phase 1 and 2 studies — 125 mg dose of palbociclib. Formulation used in phase 1 and 2 studies
Drug: Palbociclib capsule: phase 3 studies — 125 mg dose of palbociclib. Formulation used in phase 3 studies
Drug: Palbociclib capsule: ICH — 125 mg dose of palbociclib. Intended final market formulation

SUMMARY:
This study is intended to establish the equivalence of 2 formulations to the intended final market product. The formulations to compare are the capsule given to patients in the phase I and II studies and the capsule that is being administered to the patients in the phase III trials. Both capsules will be compared to the intended final market capsule. The comparison will be performed looking at the pharmacokinetic parameters that define the rate and extent of absorption, those are Cmax and AUC. A statistical analysis will be performed comparing these parameters calculated after a single 125 mg dose of the 3 capsules identifying like that if there are significant differences between these 3 formulations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or female subjects of non-childbearing potential between the ages of 18 and 55 years
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Any condition possibly affecting drug absorption

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 7 days
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 7 days

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 7 days
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 7 days
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Area Under the Curve From Time Zero to 72 hrs [AUC (0-72)] | 3 days
  AUC (0-72)= Area under the plasma concentration versus time curve from time zero (pre-dose) to 72 hrs(0-72)
Apparent Oral Clearance (CL/F) | 7 days
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Plasma Decay Half-Life (t1/2) | 7 days
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Volume of Distribution (Vz/F) | 7 days
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481020&StudyName=A%20Study%20To%20Establish%20The%20Equivalence%20Of%202%20Palbociclib%20%28PD-0332991%29%20Formulations%20To%20The%20Intended%20Final%20Market%20Product%0A